CLINICAL TRIAL: NCT00004300
Title: Phase II Study of Stereotypes and Mental Retardation: Neurobiological Basis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: University of Florida (Other)
Responsible Party: Mark Lewis, University of Florida
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11754; UF-63394
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2006-03

CONDITIONS: Stereotyped Behavior; Mental Retardation
Keywords: mental retardation; neurologic and psychiatric disorders; rare disease; stereotyped behavior
MeSH Terms: conditions — Stereotyped Behavior; Intellectual Disability; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Bromocriptine; Sertraline

INTERVENTIONS:
Drug: bromocriptine
Drug: sertraline hydrochloride

SUMMARY:
OBJECTIVES: I. Determine differences between persons with repetitive behavior disorders and matched controls on measures of motor control relevant to basal ganglia pathophysiology.

II. Determine the efficacy of bromocriptine, a dopamine agonist, in the treatment of stereotyped behavior and related behavior disorders.

III. Determine the efficacy of sertraline hydrochloride, a selective serotonin uptake inhibitor, in the treatment of repetitive behavior disorders.

IV. Identify behavioral, environmental, and biological variables with differential drug treatment response.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Motor slowness (bradykinesia) and motor control are tested in repetitive behavior disorder patients and matched controls. Group differences reflecting alterations in basal ganglia dopamine function are compared.

Behavioral assessments are conducted on each patient by trained observers. Assessments are taken at baseline and during the maintenance phase of drug treatment described below.

The efficacy of bromocriptine in the treatment of stereotypy and self-injury is determined in a randomized, double blind, placebo controlled, crossover study extending over 20 weeks. Cohorts of 6 to 8 patients first enter into a single blind placebo phase, followed by double blind treatment with placebo or bromocriptine. The crossover manipulation entails a titration phase, a maintenance phase, then a final single blind placebo condition.

The same experimental design is used to determine the efficacy of sertraline or placebo in the treatment of stereotypy and concomitant self injury and compulsions. Duration of study is 26 weeks.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of mental retardation
* High rate of stereotyped behavior, such as concomitant self-injurious and compulsive behaviors
* No diagnosis of tardive dyskinesia or akathisia

--Prior/Concurrent Therapy--

* No exposure to neuroleptics within 6 months prior to study

--Patient Characteristics--

* Age: 18 to 55
* Hematopoietic: (for bromocriptine and sertraline treatments) No history of anemia No clinically significant hematologic disease
* Hepatic: (for bromocriptine and sertraline treatments) No history of hepatic abnormalities No clinically significant liver disease
* Renal: (for bromocriptine and sertraline treatments) No history of renal abnormalities No clinically significant renal disease
* Cardiovascular: (for bromocriptine and sertraline treatments) No history of hypertension No clinically significant cardiac disease
* Other: No history of seizure within 4 months prior to study (for bromocriptine and sertraline treatments) No history of sensitivity to ergot alkaloids (for bromocriptine treatment) No sensitivity to serotonin uptake inhibitors (for sertraline treatment) No patients with sensory deficits (for motor function assessments)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Overall Officials: Mark H. Lewis, Study Chair — University of Florida
Locations (1):
- Western Carolina Center, Morganton, North Carolina, United States